CLINICAL TRIAL: NCT00097188
Title: A Phase II, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Rituximab (Mabthera/Rituxan) in Adults With Relapsing Remitting Multiple Sclerosis
Brief Title: A Study to Evaluate Rituximab in Adults With Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: U2787g
Record Dates: First submitted 2004-11-18; First posted 2004-11-19 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing remitting multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
This is a Phase II, randomized, double-blind, parallel group, placebo controlled, multicenter study to evaluate the safety and efficacy of Rituximab in adults with RRMS.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and to comply with the schedule of protocol assessments
* Age 18--55 years, inclusive
* Diagnosis of relapsing MS, as defined by McDonald Criteria 1--4
* History of at least one relapse in the subject's medical records during the 1 year prior to randomization
* EDSS at screening between 0 and 5.0 points, inclusive
* For subjects of reproductive potential (males and females), ability and willingness to use a reliable means of contraception (e.g., hormonal contraceptive, patch, vaginal ring, intrauterine device, physical barrier) during the study, including the safety follow-up period, and for up to 1 year after their last dose of study drug, even if they have discontinued early from the study

Exclusion Criteria:

* Pregnancy or lactation
* Incompatibility with MRI
* Lack of peripheral venous access
* History of severe, allergic, or anaphylactic reactions to humanized or murine monoclonal antibodies
* Known active bacterial, viral, fungal, or mycobacterial infection, or other infection (including atypical mycobacterial disease, but excluding fungal infections of nail beds or recurrent herpes infections), or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 30 days prior to screening or oral antibiotics within 14 days prior to screening
* History or presence of recurrent or chronic infection (e.g., hepatitis B or C, HIV, or syphilis)
* History of cancer, including solid tumors and hematologic malignancies (except fully resolved and resected cutaneous basal cell and squamous cell carcinomas of the skin)
* History of alcohol or drug abuse within 6 months prior to screening
* History of or currently active primary or secondary immunodeficiency
* Presence of significant, uncontrolled disease of the cardiovascular, pulmonary, renal, hepatic, endocrine, or gastrointestinal systems
* Diagnosis of secondary progressive, primary progressive, or progressive relapsing MS
* History or presence of vascular disease potentially affecting brain or spinal cord (e.g., stroke, transient ischemic attack, severe carotid stenosis, aortic aneurysm, intracranial aneurysm, hemorrhage, arteriovenous malformation)
* History or presence of myelopathy due to spinal cord compression by disk or vertebral disease
* History of severe, clinically significant CNS trauma (e.g., cerebral contusion, spinal cord compression)
* History of intracranial or intraspinal tumor (e.g., meningioma, glioma)
* History or presence of potential metabolic cause of encephalopathy or myelopathy (e.g., untreated vitamin B12 deficiency, untreated thyroid deficiency)
* History or presence of infectious causes of encephalopathy or myelopathy (e.g., syphilis, Lyme disease, human T-cell lymphotropic virus type 1 [HTLV-1], herpes zoster myelopathy)
* Neuromyelitis optica
* History or presence of systemic autoimmune disorders potentially causing progressive neurologic disease (e.g., lupus, antiphospholipid antibody syndrome, Sjogren�s syndrome, Behcet disease)
* History or presence of sarcoidosis
* Relapse within 30 days prior to randomization
* Previous treatment with rituximab (MabThera(R)/Rituxan(R))
* Treatment with any investigational agent within 90 days of randomization or five half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 30 days prior to randomization
* Previous treatment with lymphocyte-depleting therapies (e.g., Campath(R), anti-CD4, cladribine, total body irradiation, bone marrow transplantation)
* Treatment with cyclophosphamide or mitoxantrone within 12 months of randomization
* Systemic corticosteroid therapy within 30 days of randomization
* Treatment with IFN-Beta; or Copaxone(R) within 60 days of randomization
* Treatment with IVIG within 60 days of randomization
* Plasmapheresis within 60 days of randomization
* Treatment with non-lymphocyte depleting immunosuppressive therapies (e.g., azathioprine, mycophenolate mofetil, cyclosporine) within 90 days prior to randomization
* Statins or hormone replacement therapy started within 30 days of randomization
* Positive pregnancy test
* B-cell count <1.1% (reported as percent CD19)
* Vitamin B12 below the lower limit of normal with an abnormal methylmalonic acid level
* Positive rapid plasma reagin
* Serum creatinine >1.4 mg/dL for women or >1.6 mg/dL for men
* Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) >2.5 x the upper limit of normal
* Platelet count <100,000/mL
* Hemoglobin <8.5 g/dL
* Neutrophils <1.5 x 10^3/mL
* Serum IgG levels below 5.65 mg/mL and serum IgM levels below 0.55 mg/mL
* Findings on brain MRI scan consistent with clinically significant conditions other than MS
* Electrocardiogram (ECG) showing significant abnormality that the treating investigator determines may jeopardize the subject's health (i.e., acute ischemia, left bundle branch, or bifascicular block)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2004-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of rituximab compared with placebo, as measured by MRI scans of the brain for the total number of lesions observed, and to evaluate the safety and tolerability of rituximab in subjects with RRMS.

SECONDARY OUTCOMES:
To evaluate the efficacy of rituximab compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Smith, M.D., Study Director — Genentech, Inc.
Locations (31):
- United States (31):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - Loma Linda University, Loma Linda, California
  - Sutter Gould Medical Foundation, Modesto, California
  - University Of California At Davis, Sacramento, California
  - Neurological Research Institute Of East Bay, Walnut Creek, California
  - Neurology Associates, P.A., Maitland, Florida
  - Multiple Sclerosis Center of Brevard, Melbourne, Florida
  - Neurological Services Of Orlando, Orlando, Florida
  - Neurological Associates, Pompano Beach, Florida
  - MS Center of Vero Beach, Vero Beach, Florida
  - MS Center Of Atlanta, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Kentucky Neuroscience Research, Louisville, Kentucky
  - University of Maryland Hospital MS Center, Baltimore, Maryland
  - Michigan Institute For Neurological Disorders, Farmington Hills, Michigan
  - Deaconess Billings Clinical Research Division, Billings, Montana
  - Albany Medical Center, Albany, New York
  - Meritcare Neuroscience Clinic, Fargo, North Dakota
  - Neurology and Neuroscience Assoc.,INC, Akron, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - University Of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Neurology Specialists of Dallas, PA, Dallas, Texas
  - Maxine Mesinger MS Clinic/ Baylor College of Medicine, Houston, Texas
  - Neurology Clinic of San Antonio, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Holy Family MS Center, Spokane, Washington
  - Neurology and Neurosurgery Associates of Tacoma, Inc., P.S., Tacoma, Washington
  - St. Luke's Medical Center/Center for Neurological Disorders, Milwaukee, Wisconsin

REFERENCES:
- [Result] Hauser SL, Waubant E, Arnold DL, Vollmer T, Antel J, Fox RJ, Bar-Or A, Panzara M, Sarkar N, Agarwal S, Langer-Gould A, Smith CH; HERMES Trial Group. B-cell depletion with rituximab in relapsing-remitting multiple sclerosis. N Engl J Med. 2008 Feb 14;358(7):676-88. doi: 10.1056/NEJMoa0706383. PMID 18272891
- [Result] Smith CH, Waubant E, Langer-Gould A. Absence of neuromyelitis optica IgG antibody in an active relapsing-remitting multiple sclerosis population. J Neuroophthalmol. 2009 Jun;29(2):104-6. doi: 10.1097/WNO.0b013e3181a63606. PMID 19491632